CLINICAL TRIAL: NCT00744276
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Multicenter Evaluation of the Use of Topically Administered Danazol Versus Placebo in Subjects With Pain Associated With Fibrocystic Breast Disease
Brief Title: A Study of Topical Danazol for the Treatment of Pain Associated With Fibrocystic Breast Disease
Acronym: FP1198-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FemmePharma Global Healthcare, Inc. (Industry)
Responsible Party: Peter K. Mays, Ph.D. / Vice President, Pharmaceutical Development, FemmePharma Global Healthcare, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FP1198-001
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Fibrocystic Disease of Breast
Keywords: fibrocystic breast disease; fibrocystic disease of breast; breast pain; mastalgia; cyclic mastalgia; cystic breast disease
MeSH Terms: conditions — Fibrocystic Breast Disease; Mastodynia | interventions — Danazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Active Comparator)
  Interventions: Drug: danazol
- 2 (Active Comparator)
  Interventions: Drug: danazol
- 3 (Active Comparator)
  Interventions: Drug: danazol
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo
- 6 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: danazol — danazol applied topically once per day for 4 treatment cycles
  Arms: 1; 2; 3
Drug: Placebo — placebo topically applied once daily for 4 treatment cycles
  Arms: 4; 5; 6

SUMMARY:
The purpose of this study is to determine the safety of three doses of topically applied danazol compared to placebo in subjects with pain associated with fibrocystic breast disease and to determine the appropriate clinical dose for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Menstruating females at least 18 years of age
* Has moderate to severe breast pain associated with cyclical fibrocystic breast disease
* Is in good general health

Exclusion Criteria:

* Pregnant within the past 6 months or lactating
* History of malignancy or currently being treated for cancer of the breast or genital organs
* Has taken within the past 3 months or is currently taking hormonal contraception
* Has any condition for which an androgen or steroid is contraindicated
* Has had breast implants or breast reduction surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Subject reported breast pain as measured using a visual analog scale on the subject daily diary | 2 cycles pretreatment plus 4 cycles on treatment

SECONDARY OUTCOMES:
Physician assessment of breast nodularity at each treatment cycle visit | 2 cycles pretreatment plus 4 cycles on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter K. Mays, Ph.D., Study Director — FemmePharma Global Healthcare, Inc.
Locations (30):
- United States (30):
  - Women's Health Research, Phoenix, Arizona
  - Advanced Clinical Therapeutics, LLC, Tucson, Arizona
  - Impact Clinical Trials, Beverly Hills, California
  - Women's Health Care at Frost Street, San Diego, California
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - James A Simon, M.D., PC, Washington D.C., District of Columbia
  - Visions Clinical Research, Boynton Beach, Florida
  - Southeastern Integrated Medical, LLC, Gainsville, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Atlanta North Gynecology, PC, Roswell, Georgia
  - Women's Health Practice, Champaign, Illinois
  - Center for Women's Research, Chicago, Illinois
  - Physician's Research Group, Indianapolis, Indiana
  - Kentucky Medical Research Center, Lexington, Kentucky
  - MedVadis Research Corporation, Wellesley Hills, Massachusetts
  - Impact Clinical Trials, Las Vegas, Nevada
  - Delaware Valley OB/GYN and Infertility Group, PC, Lawrenceville, New Jersey
  - Phoenix OB-GYN Associates, Moorestown, New Jersey
  - UMDNJ Robert Wood Johnson Medica School Women's Health Institute, New Brunswick, New Jersey
  - Analgesic Development, Ltd., New York, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Southeastern Clinical Research, Chattanooga, Tennessee
  - Jackson Clinic, Jackson, Tennessee
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Seven Oaks Women's Center, San Antonio, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - Virginia Women's Center, Richmond, Virginia
  - Women's Clinical Research Center, Seattle, Washington

REFERENCES:
- [Background] Hughes LE, Mansel RE, Webster DJ. Aberrations of normal development and involution (ANDI): a new perspective on pathogenesis and nomenclature of benign breast disorders. Lancet. 1987 Dec 5;2(8571):1316-9. doi: 10.1016/s0140-6736(87)91204-9. PMID 2890912
- [Background] Panahy C, Puddefoot JR, Anderson E, Vinson GP, Berry CL, Turner MJ, Brown CL, Goode AW. Effects of danazol on incidence of progesterone and oestrogen receptors in benign breast disease. Br Med J (Clin Res Ed). 1987 Aug 22;295(6596):464-6. doi: 10.1136/bmj.295.6596.464. PMID 3117172
- [Background] Gateley CA, Mansel RE. Management of cyclical breast pain. Br J Hosp Med. 1990 May;43(5):330-2. PMID 2364227
- [Background] Barbieri RL. Danazol: molecular, endocrine, and clinical pharmacology. Prog Clin Biol Res. 1990;323:241-52. No abstract available. PMID 2406750
- [Background] Gumm R, Cunnick GH, Mokbel K. Evidence for the management of mastalgia. Curr Med Res Opin. 2004 May;20(5):681-4. doi: 10.1185/030079904125003377. PMID 15140333
- [Background] Vaidyanathan L, Barnard K, Elnicki DM. Benign breast disease: when to treat, when to reassure, when to refer. Cleve Clin J Med. 2002 May;69(5):425-32. doi: 10.3949/ccjm.69.5.425. PMID 12022387
- [Background] Sitruk-Ware R, Sterkers N, Mauvais-Jarvis P. Benign breast disease I: hormonal investigation. Obstet Gynecol. 1979 Apr;53(4):457-60. PMID 571588
- [Background] Wang DY, Fentiman IS. Epidemiology and endocrinology of benign breast disease. Breast Cancer Res Treat. 1985;6(1):5-36. doi: 10.1007/BF01806008. PMID 3902125
- [Background] Gledhill JM, Barker S, Wanless C, Hinson JP, Puddefoot JR, Panahy C, Goode AW, Vinson GP. Progesterone receptor induction by danazol in cultured cancer cells and the rat uterus. J Steroid Biochem Mol Biol. 1992 Oct;43(4):289-96. doi: 10.1016/0960-0760(92)90163-d. PMID 1390280
- See also: General breast health information — http://www.GoodBreastHealth.com